CLINICAL TRIAL: NCT06188013
Title: Proteomic Study of Plasma Exosomes in Patients With Diabetic Retinopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: wuhang2317
Record Dates: First submitted 2023-12-11; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Retinopathy
Keywords: plasma; exosome; Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- proliferative diabetic retinopathy: Age ≥18 years old；patients diagnosed with PDR by FFA
- non-proliferative diabetic retinopathy: Age ≥18 years old；patients diagnosed with NPDR by FFA
- diabetes mellitus without retinopathy: Age ≥18 years old；patients diagnosed with Diabetes Mellitus；patients weren't diagnosed with diabetic retinopathy
- health control: Age ≥18 years old；patients weren't diagnosed with Diabetes Mellitus

SUMMARY:
Objective: Explore the biomarkers related to proliferative diabetic retinopathy by analyzing the protein expression profile changes of plasma exosomes in patients with difference phases of diabetic retinopathy, and investigate potential molecular mechanisms and therapeutic targets. Methods: Enrich exosomes from plasma by column extraction method. NTA, WB and TEM were used to characterize the obtained exosomes, and exosome proteinomics was performed by chromatography⁃mass spectrometry. Corhorts: The study was divided into four groups: a healthy control group, a diabetic without diabetic retinopathy group, a non-proliferative diabetic retinopathy group, and a proliferative diabetic retinopathy group, with 6 cases in each group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers without diabetes/ Senile cataract patients without diabetes；
* Patients with diabetes who are diagnosed without DR, NPDR, and PDR by mydriatic fundus photography (or FFA)；

Exclusion Criteria:

* Patients with systemic diseases such as cancer, immune diseases, infectious diseases, and blood diseases；
* Patients with cerebral infarction, myocardial infarction and other cardiovascular and cerebrovascular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Plasma exosomal proteomics studies in patients with diabetic retinopathy should include healthy volunteers without diabetes mellitus and elderly cataract patients without diabetes mellitus; patients with systemic diseases such as cancer, immune disorders, infectious diseases, and hematological disorders, as well as patients suffering from cerebral infarcts, cardiac infarcts, and other cardiovascular diseases, are not eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
differential proteins of exosomes | December,2023-June,2024
  Exosomes were extracted and isolated from plasma, proteomics analysis of proteins in exosomes was performed to compare the number of types of changes in exosomal proteins of the four groups and to identify proteins that were up-regulated and/or down-regulated, and the relationship between the proteins and diabetic retinopathy was then analysed to look for possible mechanisms and therapeutic targets for diabetic retinopathy.

IPD SHARING:
Plan to Share IPD: Yes